CLINICAL TRIAL: NCT02683070
Title: Comparison of Pudendal Nerve Block With Ropivacaine and Intravenous Tramadol for Prevention of Catheter-related Bladder Discomfort: a Randomized Controlled Trial
Brief Title: Pudendal Nerve Block for Catheter-related Bladder Discomfort Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate Professor, West China Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PNB2015-306
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Catheter Site Discomfort
Keywords: Catheter-related bladder discomfort; Pudendal nerve block; Tramadol; Randomized controlled trial; catheter-related bladder discomfort prevention
MeSH Terms: interventions — Ropivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The PNB group (Experimental): Bilateral pudendal nerve block with 30ml of 0.33% ropivacaine (15ml for each side) will be performed after the completion of surgery before extubation.
  Interventions: Procedure: Bilateral pudendal nerve block
- The TRAM group (Active Comparator): Intravenous tramadol of 1.5mg/kg will be administrated after the completion of surgery before extubation.
  Interventions: Drug: Intravenous tramadol

INTERVENTIONS:
Procedure: Bilateral pudendal nerve block — Bilateral pudendal nerve block with 30ml of 0.33% ropivacaine (15ml for each side) after the completion of surgery before extubation
  Other Names: Ropivacaine
  Arms: The PNB group
Drug: Intravenous tramadol — Intravenous tramadol of 1.5mg/kg after the completion of surgery before extubation
  Other Names: Tramadol
  Arms: The TRAM group

SUMMARY:
Catheter-related bladder discomfort (CRBD) is not uncommon in male patients under general anesthesia, and it may cause patient agitation and exacerbated postoperative pain. In this study, the investigators will enroll male patients undergoing elective prostate surgery with urinary catheterization after anesthetic induction, and compare the efficacy of pudendal nerve block (PNB) and intravenous tramadol in prevention of CRBD.

DETAILED DESCRIPTION:
The PNB trial is an investigator-initiated, prospective, randomized controlled trial that will test the superiority of pudendal nerve block with 0.33% ropivacaine to intravenous tramadol 1.5mg/kg for CRBD prevention. A total of 94 patients undergoing elective prostate surgery at lithotomy position with urinary catheterization (16 G Fr Foley catheter) after anesthetic induction under general anesthesia will be enrolled at West China Hospital of Sichuan University. Patients will be divided randomly into two groups:

The PNB group: patients will be given bilateral pudendal nerve block with 30ml of 0.33% ropivacaine (15ml for each side) after the completion of surgery before extubation.

The TRAM group: patients will be given tramadol of 1.5mg/kg after the completion of surgery before extubation.

All patients will be evaluated by a research nurse who were blinded to the group assignments for outcomes at 0, 1, 2, 4, and 6h after patients' arrival in PACU, and after extraction of urinary catheter.

The primary outcome is the incidence of postoperative CRBD. The secondary outcomes include the severity of postoperative CRBD, postoperative tramadol requirement and number of patients with requiring postoperative tramadol, numeric rating scale (NRS) for postoperative pain, postoperative sufentanil requirement and number of patients with requiring postoperative sufentanil, postoperative side effects, and acceptance of indwelling urinary catheter after extraction of the catheter.

All primary and secondary endpoints will be analyzed on an intent-to-treat basis. Analyses are performed with the use of SPSS 18.0 software. The Student-t test is used to analyze demographic data in the two groups. The incidence of CRBD and side effects between groups are analyzed by Chi-square test, whereas the severity of CRBD (mild, moderate, and severe) is analyzed by Fisher's exact test. NRS scale is analyzed by the Mann-Whitney test. Postoperative tramadol and sufentanil requirement is analyzed by Z test, and the number of patients requiring tramadol for CRBD rescue treatment and sufentanil for postoperative pain will be analyzed with Fisher's exact test. A P value<0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18years to 75years.
* American Society of Anesthesiologists (ASA) physical status I, II, or Ⅲ.
* Undergoing elective prostate surgery at lithotomy position with urinary catheterization after anesthetic induction under general anesthesia.
* Glasgow Coma Scale (GCS) score of 15. Ability to communicate.

Exclusion Criteria:

* History of bladder dysfunction, such as over active bladder (OAB, urinary frequency: more than three times in the night or more than eight times in 24 h).
* History of bladder outflow obstruction.
* Neurogenic bladder.
* Impaired renal function.
* Coagulopathy.
* Known allergies to any anesthetic agent.
* Family history of malignant hyperthermia.
* Impairment of communication or cognition.
* Psychopathy.
* Active participation in another trial where the primary endpoint follow-up is ongoing.
* Unwillingness or inability to comply with protocol procedures.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative CRBD | 1 day
  Patients complained about postoperative CRBD

SECONDARY OUTCOMES:
The severity of postoperative CRBD | 1 day
  It's assessed according to the following scaling system: no CRBD indicates that there are no complaints of CRBD at all; mild indicates that complaints of CRBD exist only if the patient was asked about it; moderate indicates that patients complain of CRBD spontaneously; and severe indicates that CRBD causes a spontaneous behavioral response such as flailing limb, strong vocal response, or attempt to pull out the catheter.
Postoperative tramadol requirement | 1 day
  When moderate or severe CRBD is reported, intravenous tramadol 1.5mg/kg will be administered as a rescue treatment to reduce the bladder discomfort, and tramadol requirement will be recorded and compared.
Numeric rating scale (NRS) for postoperative pain. | 1 day
  Patients will be asked for evaluating pain intensity by themselves using this single 11-point numeric scale ranged between 0 to 10, where 0 represents "no pain" and 10 represents "worst imaginable pain" [17]. If the patient complains about pain with NRS greater than 4, intravenous sufentanil 5 μg will be administered as rescue analgetic treatment.
Postoperative sufentanil requirement | 1 day
  Intravenous sufentanil 5 μg will be administered as rescue analgetic treatment for postoperative pain, and sufentanil requirementwill be recorded and compared.
Incidences of postoperative side effects | 1 day
  Side effects include postoperative nausea/vomiting (PONV), dizziness, sedation, and dry mouth.
Acceptance of indwelling urinary catheter after extraction of the catheter | 1 week
  Patients will be asked to answer the question "Will you worry about urinary catheterization if you undergo another operation next time?". The answer "No" meant acceptance of indwelling urinary catheter, and the answer "Yes" meant unacceptance of indwelling urinary catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided whether to share IPD

REFERENCES:
- [Derived] Li JY, Liao R. Prevention of catheter-related bladder discomfort - pudendal nerve block with ropivacaine versus intravenous tramadol: study protocol for a randomized controlled trial. Trials. 2016 Sep 13;17(1):448. doi: 10.1186/s13063-016-1575-y. PMID 27618967